CLINICAL TRIAL: NCT05174624
Title: The Healthy Human Global Project - Hong Kong: A Community-based Cross-sectional Study on Genetic and Environmental Determinants of Immune Phenotype Variance in a Healthy Asian Population - Establishing a Path Towards Personalized Medicine
Brief Title: The Healthy Human Global Project - Hong Kong (HHGP-Hong Kong)
Status: Completed | Type: Observational
Sponsor: Centre for Immunology & Infection (Other)
Collaborators: The University of Hong Kong (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: UW21-549; HKUCTR-2959 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2021-12-01; First posted 2022-01-03 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Healthy; Immune System and Related Disorders
Keywords: Community based cross-sectional study; Observational cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, nasopharyngeal, stool, and hair samples from healthy adult donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FAMILY Cohort: This Cohort was part of a prospective population-based study in 2007, consisting of 46,001 participants in Hong Kong. It was the first large-scale programme to understand the determinants of physical, mental, and social wellbeing in Hong Kong. The Cohort has an excellent (99.8%) coverage of the neighbourhoods in Hong Kong and represents roughly 1% of all households, which enables detailed studies linking the social environment to physical and mental health.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Healthy Human Global Project-Hong Kong aims to elucidate the heritable and non-heritable factors that drive immunological variance within a healthy population in Hong Kong. By gaining a deeper understanding of these parameters, a path can be paved for personalised and precision medicine, tailored for an Asian population.

DETAILED DESCRIPTION:
The Healthy Human Global Project-Hong Kong (HHGP-Hong Kong) is built upon the Milieu Intérieur Consortium, a population-based study coordinated by the Institut Pasteur in Paris since 2011 (ClinicalTrials.gov study numbers NCT01699893 and NCT03905993). The Milieu Intérieur comprised of 1,000 healthy participants that are unrelated, and of Western European ancestry, to investigate inter-individual immunological variances by integrating intrinsic, environmental and genetic factors in innate immunity and adaptive immunity. Through the quantification of white blood cells by utilising standardised flow cytometry and correlating with sociodemographic variables, the Institut Pasteur team found that smoking, age, sex, and latent infection with cytomegalovirus, were the main non-genetic factors that affected variation in parameters of human immune cells.

The HHGP-Hong Kong will, therefore, replicate and adapt from the study design of Milieu Intérieur recruiting 1,000 healthy participants, drawn from the FAMILY Cohort, to better understand the immunological variance within the Hong Kong population. This Cohort was part of a prospective population-based study in 2007, consisting of 46,001 participants in Hong Kong. It was the first large-scale programme to understand the determinants of physical, mental, and social wellbeing in Hong Kong.

A technological platform will be developed to provide a personalized patient management strategy that takes into account individual genetics, previous infection history, resident microbiota, as well as personal lifestyle and environmental factors to define immune health.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects considered as healthy by the investigator based on medical history, clinical examination, laboratory results and ECG (blood sampling for laboratory assessments and ECG should be done at V0 and only after signed informed consent)
2. Subjects who, according to the investigator, can and will comply with the requirements of the protocol and are available for all scheduled visits at the investigational site.
3. Healthy male or female aged between 20 and 79 (included) years
4. Self-declared Han ethnicity for 3 generations
5. Body mass index (BMI) of ≥ 18.5 and ≤ 27.0 kg/m²
6. Ability to give their informed consent in writing
7. Must understand spoken Cantonese and written Chinese
8. Current participants enrolled in the FAMILY Cohort or their affiliates (i.e. any individuals referred by a FAMILY Cohort participant), or Hong Kong residents.

Exclusion Criteria:

1. Participation in the last 3 months or concurrent participation in another clinical study in which the subject has been exposed to a medical intervention including but not limited to pharmaceutical product or placebo or medical device
2. First-degree relative to previously recruited individuals in the study cohort
3. For women: pregnant or breastfeeding or intending to become pregnant or peri-menopausal

   3.1 Peri-menopausal women as defined by menstrual irregularity: either a change in the menstrual cycle length of more than seven days (early perimenopause) or two or more missed periods with an interval of 60 days or more between periods (late perimenopause)
4. Any physical exercise within the last 4 hours before inclusion (V1)
5. Subjects following a special diet for medical reasons as prescribed by a general practitioner or dietician (e.g. calorie-restricted or weight-loss diet for significant overweight, cholesterol-lowering diet or subjects suffering from any clinically diagnosed food allergy or intolerance)
6. Binge drinking (drinking at least 5 cans of beer, 5 glasses of table wines or 5 pegs of spirits on a single occasion), >2 episodes within 3 months before inclusion
7. Illicit drug use or substance abuse within 3 months before inclusion
8. Presence of evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to participate in the study satisfactorily.
9. Severe/chronic/recurrent pathological conditions, among them:

   9.1. Past or present diagnosed cancer, lymphoma, leukaemia

   9.2. Personal history of organ transplant

   9.3. Congenital or acquired immune deficiency (any confirmed or suspected immunosuppressive or immunodeficient condition, including a history of HIV infection)

   9.4. Personal history of auto-immune diseases requiring or having previously required treatment (e.g. Rheumatoid Arthritis, Systemic Lupus Erythematosus, Sarcoidosis, Ankylosing Spondylitis, Autoimmune Haemolytic Anaemia, Autoimmune Thrombocytopenic Purpura, Crohn's Disease, Psoriasis, Scleroderma, Wegener's Granulomatosis, Type I Diabetes, Thyroiditis etc.)

   9.5. Splenectomy

   9.6. Acute or chronic, clinically significant, as determined by the investigator, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests

   9.7. History of clinically significant, as determined by the investigator, neurological disorder of seizures

   9.8. Infectious diseases

   9.8.1. Chronic/ latent infection (e.g. HIV, hepatitis B virus, hepatitis C virus, HTLV, except herpes viruses such as CMV and VZV) or current acute infection or past acute infection based on investigator's judgment within the last 3 months,

   9.8.2. Presence of a rectal temperature ≥38.4°C, or axillary temperature ≥37.5°C, or intra-auricular temperature ≥38.4 °C, or buccal temperature ≥38°C on the scheduled date of inclusion,

   9.8.3. Subject receiving (currently or in the last 3 months) antibiotics, intestinal, nasal or respiratory antiseptics.

   9.9. Severe High Blood Pressure, defined as systolic BP≥160 mmHg and/or diastolic BP≥100 mmHg (2020 International Society of Hypertension Global Hypertension Practice Guidelines, grade 2 hypertension). Treated and controlled high blood pressure or documented white coat hypertension is allowed.

   9.10. Type II diabetes mellitus requiring treatment with any medication. Diabetes mellitus treated by exercise and diet control only is permitted.

   9.11. Chronic renal impairment as defined by Renal Insufficiency: glomerular filtration rate (GFR) <60 mL/min/1.73 m²16

   9.12. Chronic bone disease as treated by bisphosphonates

   9.13. Any significant disorder of coagulation or treatment with direct oral anticoagulants (DOACs) or warfarin derivatives or heparin or antiplatelet medications within 2 months preceding inclusion.

   9.14. Dermatologic conditions: any current dermatological disorder that is severe enough to prevent skin biopsy (e.g. eczema, psoriasis, acute or chronic dermatitis)

   9.15. Severe acute and chronic allergy

   9.15.1. Severe Asthma defined as asthma that is uncontrolled despite adherence with optimized high dose inhaled corticosteroid- long-acting beta2-agonist (ICS-LABA) therapy and treatment of contributory factors, or that worsens when high dose treatment is decreased,

   9.15.2. Severe food allergy, as defined by a history of giant urticaria, Quincke oedema or anaphylactic shock,

   9.15.3. Severe insect bite allergy with a history of giant urticaria, Quincke oedema or anaphylactic shock,

   9.15.4. Atopic dermatitis treated with medication.
10. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months before the inclusion. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
11. Chronic administration of NSAIDs, including aspirin: prolonged intake (> 2 weeks) within 6 months before the study or any intake [exception for low dose aspirin: maximum 250mg/daily]
12. Receipt of any vaccination 6 weeks before the inclusion or planning to receive any vaccination during the study
13. Receipt of blood products or immunoglobulins within 3 months before the inclusion or planning to receive blood products or immunoglobulins during the study
14. Haemoglobin measurement less than 10.0 g/dL for women and less than 11.5 g/dL for men
15. Platelet count less than 120.000/mm3
16. Alanine aminotransferase (ALAT) and/or aspartate transaminase (ASAT) > 3 times the upper limit of the norm (ULN)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The HHGP- Hong Kong will recruit 1,000 healthy participants, drawn from the FAMILY Cohort, its affiliates, or Hong Kong residents, to better understand the immunological variance within the Hong Kong population. This Cohort was part of a prospective population-based study in 2007, consisting of 46,001 participants in Hong Kong. It was the first large-scale programme to understand the determinants of physical, mental, and social wellbeing in Hong Kong. The Cohort has an excellent (99.8%) coverage of the neighbourhoods in Hong Kong and represents roughly 1% of all households, which enables detailed studies linking the social environment to physical and mental health.
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Factors underlying immunological variance within the general healthy population | Through study completion, an average of 1 year
  To identify factors (genetic, immunology and environmental) that contributes to the observed heterogeneity in immune responses (individual and population levels)
Naturally occurring variability of human response | Through study completion, an average of 1 year
  To characterise the naturally occurring variability of human response using whole genome sequencing and single nucleotide polymorphisms (SNPs) haplotyping
Stimulated cytokine/chemokine measurement | Through study completion, an average of 1 year
  To determine and measure cytokine/chemokine stimulated by 16 pattern-recognition receptors agonists (PRR agonists) or immune stimulators
Characterisation of commensal airway and gut microbiota | Through study completion, an average of 1 year
  To characterise commensal microbiota (nasopharyngeal swab and stool samples) in the study population
Metagenomic architecture of faecal and nasal samples | Through study completion, an average of 1 year
  To evaluate the metagenomic architecture of the population based on sequence analysis of bacterial, fungal and viral populations in faecal and nasal samples
Immune response and nutrition association | Through study completion, an average of 1 year
  To associate immune response with nutrition data
Immune phenotype variance association with genetic polymorphisms and enterotype | Through study completion, an average of 1 year
  To associate immune phenotype variance with genetic polymorphisms and enterotype
Heart rate variability with clinical and epidemiological data association | Through study completion, an average of 1 year
  To associate heart rate variability with clinical and epidemiological data
Inflammation with physical and mental health outcome association | Through study completion, an average of 1 year
  To associate inflammation with physical and mental health outcomes

SECONDARY OUTCOMES:
Genotype-to-phenotype associations at a mechanistic level | Through study completion, an average of 1 year
  To determine genotype-to-phenotype associations at a mechanistic level
Retrospective and prospective clinical and epidemiological data correlation with FAMILY Cohort | Through study completion, an average of 1 year
  To correlate retrospective and prospective clinical data with and epidemiological data from the FAMILY Cohort
Immune variation comparison between healthy European (Milieu Intérieur) and Asian (HHGP- Hong Kong) populations | Through study completion, an average of 1 year
  To compare immune variation between healthy European (Milieu Intérieur) and Asian (HHGP- Hong Kong) populations

CONTACTS AND LOCATIONS:
Overall Officials: James Di Santo, Principal Investigator — Centre for Immunology & Infection; Darragh Duffy, Principal Investigator — Centre for Immunology & Infection; Michael Ni, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Centre for Immunology & Infection Research Clinic, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided
All personal information obtained in the research project will remain strictly confidential and will not be disclosed to or seen by any person other than the authorised researchers involved. All information obtained about the participants will be stored in a locked cabinet in a security-accessible area, and also in a password-protected database at The School of Public Health, The University of Hong Kong. All personal data will be anonymised for data analysis. Data and information may be inspected by regulatory authorities of academic research, such as the Institutional Review Board of the University of Hong Kong / Hospital Authority Hong Kong West Cluster, with the accompany of research staff. Any data and sample access request from local/international researchers or collaborators must comply with regulations as elaborated by international bodies/agreements including Declaration of Helsinki.

REFERENCES:
- [Background] Delhalle S, Bode SFN, Balling R, Ollert M, He FQ. A roadmap towards personalized immunology. NPJ Syst Biol Appl. 2018 Feb 6;4:9. doi: 10.1038/s41540-017-0045-9. eCollection 2018. PMID 29423275
- [Background] Tsang JS, Schwartzberg PL, Kotliarov Y, Biancotto A, Xie Z, Germain RN, Wang E, Olnes MJ, Narayanan M, Golding H, Moir S, Dickler HB, Perl S, Cheung F; Baylor HIPC Center; CHI Consortium. Global analyses of human immune variation reveal baseline predictors of postvaccination responses. Cell. 2014 Apr 10;157(2):499-513. doi: 10.1016/j.cell.2014.03.031. PMID 24725414
- [Background] Carr EJ, Dooley J, Garcia-Perez JE, Lagou V, Lee JC, Wouters C, Meyts I, Goris A, Boeckxstaens G, Linterman MA, Liston A. The cellular composition of the human immune system is shaped by age and cohabitation. Nat Immunol. 2016 Apr;17(4):461-468. doi: 10.1038/ni.3371. Epub 2016 Feb 15. PMID 26878114
- [Background] Aziz N, Detels R, Quint JJ, Gjertson D, Ryner T, Butch AW. Biological variation of immunological blood biomarkers in healthy individuals and quality goals for biomarker tests. BMC Immunol. 2019 Sep 14;20(1):33. doi: 10.1186/s12865-019-0313-0. PMID 31521107
- [Background] Brodin P, Davis MM. Human immune system variation. Nat Rev Immunol. 2017 Jan;17(1):21-29. doi: 10.1038/nri.2016.125. Epub 2016 Dec 5. PMID 27916977
- [Background] Whitacre CC. Sex differences in autoimmune disease. Nat Immunol. 2001 Sep;2(9):777-80. doi: 10.1038/ni0901-777. No abstract available. PMID 11526384
- [Background] Thomas S, Rouilly V, Patin E, Alanio C, Dubois A, Delval C, Marquier LG, Fauchoux N, Sayegrih S, Vray M, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. The Milieu Interieur study - an integrative approach for study of human immunological variance. Clin Immunol. 2015 Apr;157(2):277-93. doi: 10.1016/j.clim.2014.12.004. Epub 2015 Jan 3. PMID 25562703
- [Background] Patin E, Hasan M, Bergstedt J, Rouilly V, Libri V, Urrutia A, Alanio C, Scepanovic P, Hammer C, Jonsson F, Beitz B, Quach H, Lim YW, Hunkapiller J, Zepeda M, Green C, Piasecka B, Leloup C, Rogge L, Huetz F, Peguillet I, Lantz O, Fontes M, Di Santo JP, Thomas S, Fellay J, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Natural variation in the parameters of innate immune cells is preferentially driven by genetic factors. Nat Immunol. 2018 Mar;19(3):302-314. doi: 10.1038/s41590-018-0049-7. Epub 2018 Feb 23. PMID 29476184
- See also: HKU Clinical Trials Registry website — http://www.hkuctr.com/Study/Show/a3831f8f1e674e8f90eb3d8e12958a02